CLINICAL TRIAL: NCT05364372
Title: Symptom Management and Lifestyle Intervention With Hispanic Cancer Survivors and Caregivers
Brief Title: SMLI With Hispanic Cancer Survivors and Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 35221
Record Dates: First submitted 2022-04-29; First posted 2022-05-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cancer Survivors; Cancer
Keywords: Cancer survivors; Caregivers; Symptom assessment; Lifestyle intervention; Diet; Physical activity
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Attention control (Active Comparator): Dyads will receive mailed print education materials regarding healthy lifestyle (nutrition and physical activity) disseminated by ACS and NCI. They will also receive 12 weekly phone calls to assess post-treatment related symptoms.
  Interventions: Behavioral: Symptom assessment only
- Symptom management and lifestyle intervention (Experimental): Dyads will receive 12 weekly telephone-based coaching sessions, a participant educational handbook, and a pedometer for self-monitoring physical activity.
  Interventions: Behavioral: Symptom management and lifestyle intervention

INTERVENTIONS:
Behavioral: Symptom assessment only — Dyads will receive 12 weekly phone calls to assess symptom management.
  Arms: Attention control
Behavioral: Symptom management and lifestyle intervention — Survivor and caregiver dyads will work together with a coach to establish diet and physical activity change SMART goals. Motivational interviewing based weekly coaching sessions will review symptom management and goal attainment and then enact strategies to modify goals to be more relevant and achievable.
  Arms: Symptom management and lifestyle intervention

SUMMARY:
Fewer than 20% of Hispanic cancer survivors meet the American Cancer Society's (ACS) Guidelines on Nutrition and Physical Activity. Diagnosed at younger ages, later stages and with fewer resources (e.g., access to care), Hispanic cancer survivors are more likely to suffer from many symptoms, which linger long after they have completed treatment and may prevent them from leading a healthy life. Healthier lifestyle behaviors (such as diet and physical activity) would result in an immediate benefit of reduced symptoms and long-term benefit of improved health while lowering cancer risk. This randomized controlled trial tests an intervention that will help in lessening survivors' symptoms to improve adherence to the ACS guidelines for cancer prevention ultimately improving overall health.

DETAILED DESCRIPTION:
In the proposed randomized controlled trial, the investigators will test the 12-week SMLI against an attention control condition in 107 dyads of Hispanic cancer survivors who have completed curative treatments within the past two years and their informal caregivers. A 12-week follow-up will determine the sustainability of the intervention. The primary outcome of this trial, vegetable and fruit intake in survivors (secondary in caregivers), will be measured at baseline, 13, and 25 weeks, using validated methods. Additional secondary and exploratory outcomes will add to the rigor of the trial and provide robust findings for future dissemination efforts.

Specific Aim #1: Test the efficacy of the SMLI as compared to attention control among Hispanic female cancer survivors and their caregivers with respect to:

1. Increase in fruit and vegetable consumption (measured via self-reported 24-hour recall and objectively with carotenoid skin colorimetry)
2. Increase in physical activity (Metabolic Equivalents hours/week of moderate to vigorous physical activity measured by actigraphy) and decrease in symptom severity index

Specific Aim #2: Determine the extent to which improvements in primary and secondary outcomes over weeks 13 and 25 are mediated by social support and self-efficacy.

ELIGIBILITY:
Inclusion criteria for female Hispanic cancer survivors:

1. 18 years of age or older;
2. have access to a telephone,
3. speak and understand English or Spanish;
4. have finished curative intent treatment for cancer within the previous 10 years and do not have any subsequent cancer treatments planned, except for non-curative intent maintenance therapy, such as hormonal therapy;
5. must have at least 1 of the 5 most common cancer-related symptoms (pain, sleep disturbance, anxiety, depression and/or fatigue) with a severity score of 4 or higher on a 0-10 rating scale (based on NCCN guidelines for symptom monitoring and management used successfully in past work); and
6. has a caregiver willing to participate in the study with them.

Inclusion criteria for the caregivers (nominated by the survivor) are:

1. age 18 or older;
2. able to speak and understand English or Spanish;
3. access to a telephone; and
4. not currently treated for cancer preserving the distinction between survivor and caregiver. The caregiver can be of any race or ethnicity and any gender.

Exclusion criteria for survivors:

1. Under the age of 18 years
2. Does not have access to a telephone
3. Completed treatment for cancer more than 1 year ago
4. Currently receiving counseling or treatment for special diet or weight loss
5. Does not have a caregiver willing to participate with them

Exclusion criteria for caregivers:

1. Under the age of 18 years
2. Does not have access to a telephone
3. Currently receiving counseling or treatment for special diet or weight loss
4. Currently being treated for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 217 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in vegetable and fruit intake at 13-weeks in survivors | Baseline to 13-weeks
  Measured using data from 24-hour dietary recalls conducted on three randomly chosen days per timepoint including one weekend day and two weekdays. Objective assessment will be conducted in 10% of the sample using the Veggie Meter® Skin Carotenoid Scanner which measures skin carotenoid levels.
Change from baseline vegetable and fruit intake at 25-weeks in survivors | Baseline to 25-weeks
  Measured using data from 24-hour dietary recalls conducted on three randomly chosen days per timepoint including one weekend day and two weekdays. Objective assessment will be conducted in 10% of the sample using the Veggie Meter® Skin Carotenoid Scanner which measures skin carotenoid levels.

SECONDARY OUTCOMES:
Physical activity | Baseline, 13-weeks, and 25-weeks
  Objective measurement will be completed using an Actigraph GTX9 accelerometer which participants will be mailed and then instructed to wear on the hip for seven continuous days. From the Actigraph GTX9 we get daily minutes of moderate to vigorous physical activity, sleep, sedentary time, light physical activity, and steps taken. Averages over 5-7 days will be used for physical activity measures (daily minutes of activity) to ensure validity and reliability. Participants will also provide a self-report using a seven day recall of physical activity.
Symptom severity | Baseline, 13-weeks, and 25-weeks
  The General Symptom Distress Scale will be used to evaluate 12 symptoms: shortness of breath, pain, sleep difficulties, diarrhea, constipation, numbness or tingling, swelling in hands and feet, difficulty concentrating, poor appetite, depression, anxiety, fatigue. Respondents indicate presence of each symptom (yes/no) and rate its severity on the scale from 1 to 10.
Vegetable and fruit intake in caregivers | Baseline, 13-weeks, and 25-weeks
  Measured using data from 24-hour dietary recalls conducted on three randomly chosen days per timepoint including one weekend day and two weekdays. Objective assessment will be conducted in 10% of the sample using the Veggie Meter® Skin Carotenoid Scanner which measures skin carotenoid levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bea, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No